CLINICAL TRIAL: NCT03800368
Title: 12-week Aerobic-Anaerobic Transition Exercise Intervention and Overnight Sleep-dependent Procedural Memory Consolidation in Patients With Schizophrenia
Brief Title: Exercise and Overnight Motor Sequence Task
Acronym: EOMST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Lincoln Lik-Hang Lo, Postdoctoral Fellow, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HKU_Psych
Record Dates: First submitted 2019-01-03; First posted 2019-01-11 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Schizophrenia and Related Disorders; Psychotic Disorders
Keywords: Exercise; Sleep-dependent memory consolidation; Aerobic; Anaerobic
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-endurance group (Experimental): This group of subjects will receive 2-3 sessions of high-intensity cycling exercise training per week, for a total of 12 weeks. The exercise the subjects received will interchange between the aerobic and anaerobic state.
  Interventions: Other: Exercise
- Low-endurance group (Experimental): This group of subjects will receive 2-3 sessions of low-intensity cycling exercise training per week, for a total of 12 weeks. The exercise the subjects received will maintain at an aerobic level.
  Interventions: Other: Exercise
- Psycho-education (Active Comparator): This group of subjects will receive 2-3 sessions of psycho-education class per week, for a total of 12 weeks. The content of the class includes non-exercise related psycho-education content to participants (e.g., food hygiene, psychological well being, food nutrition, etc).
  Interventions: Other: Non-exercise

INTERVENTIONS:
Other: Exercise — Indoor cycling exercise intervention
  Arms: High-endurance group; Low-endurance group
Other: Non-exercise — Psycho-education
  Arms: Psycho-education

SUMMARY:
The objective of this randomized controlled trial (RCT) is to compare the changes of the sleep-related memory functions in patients with psychosis after they have completed the 12-week high-intensity exercise intervention, the 12-week low-intensity exercise intervention, or the 12-week controlled non-exercise intervention respectively. Fifty-one patients with psychosis, patients who received either the high-intensity exercise or low-intensity exercise as intervention shown a significant improvement to their impaired sleep-related memory function, while those who received non-exercise intervention has no such improvement. Moreover, high-intensity exercise may have a more prominent effect compare to low-intensity exercise.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 55
* Based on the SCID diagnosed to have schizophrenia and related psychotic disorders
* Ability to understand the nature of the study and to give written informed consent

Exclusion Criteria:

* Severe physical illness (Myocardial Infarction, Hypertension, Fracture, Spinal problems in which exercise may be contraindicated), and seizure disorders
* Comorbid substance dependence
* Unstable psychotic symptoms
* A history of brain trauma or organic brain disease
* Known history of intellectual disability or special school attendance
* Answered one or more "yes" in the PAR-Q and without doctors approval for exercise

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2016-12-21 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
The sleep-dependent procedural memory consolidation after 12 weeks of intervention | 12-week Follow-up
  Tested by comparing the finger-tapping motor sequence task performance between the three groups during the 12-week follow-up assessment.

SECONDARY OUTCOMES:
The verbal memory consolidation after 12 weeks of intervention | 12-week Follow-up
  Tested by comparing the logical memory task performance between the three groups during the 12-week follow-up assessment
The attention performance after 12 weeks of intervention | 12-week Follow-up
  Measured by using the cancellation task performance and compare between the three groups during the 12-week follow-up assessment
The sleep quality after 12 weeks of intervention | 12-week Follow-up
  Measured by using the Pittsburgh Sleep Quality Index (PSQI) and compare the differences between the three groups during the 12-week follow-up assessment
The insomnia severity after 12 weeks of intervention | 12-week Follow-up
  Measured by using the Insomnia Severity Index (ISI) and compare the differences between the three groups during the 12-week follow-up assessment

CONTACTS AND LOCATIONS:
Overall Officials: Lik Hang Lincoln Lo, Principal Investigator — The University of Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lo LLH, Lee EHM, Hui CLM, Chong CSY, Chang WC, Chan SKW, Lin JJ, Lo WTL, Chen EYH. Effect of high-endurance exercise intervention on sleep-dependent procedural memory consolidation in individuals with schizophrenia: a randomized controlled trial. Psychol Med. 2023 Apr;53(5):1708-1720. doi: 10.1017/S0033291721003196. Epub 2021 Oct 7. PMID 34615565